CLINICAL TRIAL: NCT05366777
Title: Effect of an Intravenous Acetaminophen/Ibuprofen Fixed-dose Combination on Postoperative Opioid Consumption and Pain After Video-assisted Thoracic Surgery: A Double-blind Randomized Controlled Trial
Brief Title: Intravenous Acetaminophen/Ibuprofen Fixed-dose Combination on Postoperative Opioid Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Kyongbo Pharmaceutical (Unknown)
Responsible Party: Principal Investigator, Hojin Lee, MD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Maxigesic_Lung
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Postoperative Pain
Keywords: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Ibuprofen; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A prospective randomized double-blinded study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The nurse who is not involved in this study knows the allocated group and sends the bottle of the drug which looks the same in both groups, to the operation room and ward.
  The care provider, investigator, patients, and outcomes assessor will be not informed of the infusion of the drug by not attaching an identifiable label so that it cannot be distinguished from normal saline.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maxigesic group (Experimental): At the end of induction, the Maxigesic group will receive intravenous acetaminophen (1000 mg)/ibuprofen (300 mg) for 15 min, every 6 hours, a total of 4 times.
  Interventions: Drug: acetaminophen/ibuprofen fixed-dose combination
- Control group (Placebo Comparator): At the end of induction, the control group will receive intravenous normal saline with the same volume and same time points as the intervention group receives.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: acetaminophen/ibuprofen fixed-dose combination — Intravenous acetaminophen (1000 mg)/ibuprofen (300 mg) fixed-dose combination (total 100 ml)
  Other Names: Maxigesic
  Arms: Maxigesic group
Drug: Saline — 100 ml of normal saline
  Other Names: Placebo
  Arms: Control group

SUMMARY:
This prospective, randomized, double-blinded study is designed to evaluate the postoperative analgesic effect of the intravenous acetaminophen/ibuprofen fixed-dose combination in patients undergoing video-assisted thoracic surgery (VATS). We hypothesize that the intravenous acetaminophen/ibuprofen fixed-dose combination can significantly reduce postoperative opioid consumption and pain severity in patients with VATS.

DETAILED DESCRIPTION:
Adult patients undergoing elective unilateral VATS wedge resection, segmentectomy, or lobectomy are randomly allocated to receive intravenous acetaminophen (1000 mg)/ibuprofen (300 mg) fixed-dose combination (n=48) or not (n=48). At the end of induction, the intervention group will receive intravenous acetaminophen (1000 mg)/ibuprofen (300 mg) for 15 min, every 6 hours, a total of 4 times. The control group will receive intravenous normal saline with the same volume and same time points as the intervention group receives.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective unilateral VATS segmentectomy or lobectomy under general anesthesia
* American Society of Anesthesiologists (ASA)physical classification I-II
* Consent to IV-patient controlled analgesia use
* Willingness and ability to sign an informed consent document

Exclusion Criteria:

* Do not understand our study
* Allergies to anesthetic or analgesic medications
* Continuous local anesthetics infiltration for postoperative pain control
* Patients who receive mechanical ventilation more than 2 hours after surgery
* Pregnancy/Breastfeeder
* Medical or psychological disease that can affect thetreatment response

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Total fentanyl consumption during 24 hours | postoperative 24 hours
  postoperative fentanyl consumption (mcg) via IV patient controlled analgesia

SECONDARY OUTCOMES:
Total fentanyl consumption | postoperative 6, 48 hours
  postoperative fentanyl consumption (mcg) via IV patient controlled analgesia
Postoperative pain score | postoperative 6, 24, 48 hours
  11-pointed NRS pain score at resting/coughing NRS (0-10): 0,"no pain"; 10, "worst pain imaginable"
Postoperative nausea and vomiting | postoperative 24, 48 hours
  Incidence of postoperative nausea and vomiting (%)
Quality of recovery-15 | postoperative 24, 48 hours
  Korean version of Quality of recovery-15 questionnaire (0-150): 0, "very poor recovery"; 150, "excellent recovery"

CONTACTS AND LOCATIONS:
Overall Officials: Hojin Lee, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided